CLINICAL TRIAL: NCT03685838
Title: A Randomised Controlled Trial of Compression Stockings Therapy Following Mechano-Chemical Ablation
Brief Title: Compression Stockings Therapy Following Mechano-Chemical Ablation (Clarivein®)
Acronym: COMMOCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMMOCA
Record Dates: First submitted 2018-09-21; First posted 2018-09-26 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Varicose Veins; Chronic Venous Insufficiency
Keywords: mechano-chemical ablation; compression stockings
MeSH Terms: conditions — Varicose Veins | interventions — Stockings, Compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression (Active Comparator): Patient will receive Class II above knee compression stockings, and will be asked to wear it for 1 week. This would involve wearing the stocking during daytime but patients will be allowed to take it off at night whilst in bed.
  Interventions: Other: Compression Stockings
- No Compression (No Intervention): Patient will not receive any compression stockings.

INTERVENTIONS:
Other: Compression Stockings — Class II above knee compression stockings
  Arms: Compression

SUMMARY:
This study will be looking at the effect of compression therapy in patients having Mechano-Chemical Ablation (MOCA) therapy for truncal incompetence of their varicose veins using the ClariVein® device. Patients will be randomised to either the compression group (group A) or the no compression group (group B).

The pain scores, compliance, quality of life scores, occlusion rate at 6 months as well as the cost effectiveness of each intervention will be assessed.

DETAILED DESCRIPTION:
Varicose veins are common and are known to affect approximately one third of the population. Chronic Venous Disease (CVD) has been shown to have a negative impact on the quality of life of patients and treatment of varicose veins has been demonstrated to lead to improvement in the quality of life of patients. Over the past decade, new endovenous techniques have been introduced and these are felt to be cost-effective, especially, when performed in an outpatient or 'office-based' setting.

There is currently uncertainty about the use of compression stockings following treatment of varicose veins. International Union of Phlebology (IUP), The Society for Vascular Surgery and the American Venous Forum, as well as 2013 National Institute for Health and Care Excellence (NICE) Guideline on Varicose Veins in the Legs have recommended that compression stockings are suitable in certain clinical indications and can be worn post-operatively for no more than 7 days after interventional treatment to prevent haematoma formation, pain and swelling. However, further research is essential for determining clinical and cost effectiveness, as well as length of time compression should be worn, and level of compression.

Several researchers have looked into the practice of using compression after venous ablation. In a survey of the management of varicose veins by the members of the Vascular Society of Great Britain and Ireland. Edwards et al. found that the majority of surgeons used bandages post-operatively, with 49% using elastic bandage. To date, the literature on the use of compression stockings following treatment of varicose veins is limited.

Mechano-Chemical Ablation (MOCA) combines mechanical damage to the endothelium caused by a rotating wire with simultaneous catheter-guided infusion of a liquid sclerosant that irreversibly damages the cellular membrane of the endothelium, causing fibrosis of the vein. The exact mechanism is still not exactly known. However, recent experimental research showed that various sclerosants induced apoptosis in the vein wall rather than having an effect restricted to the endothelium. Incomplete loss of endothelial cells and penetration of the sclerosant effect into the media suggest that medial damage is crucial to the success of sclerotherapy and may explain why it is less effective in larger veins. This poses the question whether compression is needed post sclerotherapy to improve contact of the sclerosant to the endothelium when media penetration seems to be more important to allow apoptosis of smooth muscle cells.

The investigators therefore propose to undertake a randomised study looking at the effect of compression therapy after MOCA using Clarivein device

ELIGIBILITY:
Inclusion Criteria:

* Age>=21 to <=80
* Able to walk unassisted and attend follow-up visits
* Symptomatic Great Saphenous Vein (GSV) or Small Saphenous Vein (SSV) vein reflux >0.5 seconds on colour Duplex ultrasound
* Able to provide informed consent

Exclusion Criteria:

* Previous or current deep vein thrombosis or pulmonary embolism
* Patients with a hypercoaguable state
* Previous thrombophlebitis in the truncal vein in question, which had recanalized and was now incompetent on duplex ultrasound
* Recurrent varicose vein i.e. patients who have had treatment previously in the designated truncal vein with any modality
* Patients who have had treatment in either leg for an incompetent saphenous truncal vein less than 3 months prior to treatment and enrolment into this study
* Patients requiring adjuvant treatment of varicose veins
* Arterial disease (ABPI < 0.6 and the absence of a palpable pedal pulse)
* Vein diameter <3mm or >12mm as measured in the standing position on duplex ultrasound
* Varicose veins unsuitable for MOCA (e.g. very tortuous vein)
* Pregnancy
* Lycra, sclerosant or local anaesthetic allergy
* Patients who have opted for an alternative method of treatment
* Patients with fibromyalgia
* Patients with Clinical, Etiologic, Anatomic and Pathophysiologic (CEAP) score of C6 (active ulcer), C1 and C2 (asymptomatic) disease
* Patients with a life expectancy less than 12 months
* Inability or unwillingness to complete questionnaires
* Patients who refuses to participate and unable to provide informed consent or comply with the study protocol.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-02-13 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain Score post-procedure | First 10 days post-procedure
  Participants will record their pain score using the Visual Analogue Score (VAS) for pain. The scale ranges from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Quality of Life score using the EQ-5D questionnaire | Baseline, 2 weeks post-op, 6 months post-op
  EQ-5D is used to assess quality of life based on Mobility, Self-care, Usual Activities, Pain/Discomfort and Anxiety, rated at 5 levels: no problems, slight problems, moderate problems, severe problems, unable to perform activity. Inputs from this questionnaire is used to observe for changes in quality of life overtime
Quality of life score using the Chronic Venous Insufficiency Questionnaire (CIVIQ) | Baseline, 2 weeks post-op, 6 months post-op
  CIVIQ-14 is a questionnaire based on three dimensions - pain, physical and psychological, based on a scale from 1 to 5 (no trouble, slight, moderate, considerable, severe). Based on inputs, Global Index Score (GIS) will be tabulated, ranging from 0 to 100 - the higher the value, the poorer the quality of life.
Quality of life score using the Aberdeen Varicose Veins Questionnaire (AVVQ) | Baseline, 2 weeks post-op, 6 months post-op
  To measure health status of varicose vein patients based on symptoms and impact on daily activities. A total score ranging from 0 to 100 will be tabulated, with 100 being worst quality of life
Clinical Change using Venous Clinical Severity Score (VCSS) | Baseline, 2 weeks post-op, 6 months post-op
  VCSS evaluates the severity of hallmarks of venous disease - 0 (none), 1 (Mild) , 2(Moderate), 3 (Severe).
Time taken to return to work and normal activities | 10 days post-op
Degree of bruising and phlebitis | 2 weeks post-op, 6 months post-op
  Assessed using a pre-determined score (0=0%; 1= <25% of treated vein affected; 2 = 25-50% ; 3 = 50-75%; 4 = 75-100% and 5 = extending beyond the treated vein
The number of patient compliant with the intervention | 10 days post-op
Patient's satisfaction | 2 weeks post-op, 6 months post-op
  To rate satisfaction with overall teatment regime with a numerical scale of 0 (least satisfied) to 10 (most satisfied)
Comparison of the cost-effectiveness of the intervention | 6 months post-op
  Analyze cost and patient outcomes to determine effectiveness of interventions
Successful obliteration of target vein | 2 weeks post-op, 6 months post-op
  This is assessed by duplex ultrasound scan. Recanalization will be defined by a segment of vein greater than or equal to 5cm

CONTACTS AND LOCATIONS:
Overall Officials: Tang Tjun Yip, Principal Investigator — Singapore General Hospital
Locations (2):
- Galway University Hospital, Galway, Galway, Ireland
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans CJ, Fowkes FG, Ruckley CV, Lee AJ. Prevalence of varicose veins and chronic venous insufficiency in men and women in the general population: Edinburgh Vein Study. J Epidemiol Community Health. 1999 Mar;53(3):149-53. doi: 10.1136/jech.53.3.149. PMID 10396491
- [Background] Sakurai H, Naito H. A cross-resistance of Pyricularia oryzae Cavara to kasugamycin and blasticidin S. J Antibiot (Tokyo). 1976 Dec;29(12):1341-2. doi: 10.7164/antibiotics.29.1341. No abstract available. PMID 1051420
- [Background] Biemans AA, Kockaert M, Akkersdijk GP, van den Bos RR, de Maeseneer MG, Cuypers P, Stijnen T, Neumann MH, Nijsten T. Comparing endovenous laser ablation, foam sclerotherapy, and conventional surgery for great saphenous varicose veins. J Vasc Surg. 2013 Sep;58(3):727-34.e1. doi: 10.1016/j.jvs.2012.12.074. Epub 2013 Jun 13. PMID 23769603
- [Background] MacKenzie RK, Paisley A, Allan PL, Lee AJ, Ruckley CV, Bradbury AW. The effect of long saphenous vein stripping on quality of life. J Vasc Surg. 2002 Jun;35(6):1197-203. doi: 10.1067/mva.2002.121985. PMID 12042731
- [Background] van den Bos R, Arends L, Kockaert M, Neumann M, Nijsten T. Endovenous therapies of lower extremity varicosities: a meta-analysis. J Vasc Surg. 2009 Jan;49(1):230-9. doi: 10.1016/j.jvs.2008.06.030. Epub 2008 Aug 9. PMID 18692348
- [Background] Gloviczki P, Comerota AJ, Dalsing MC, Eklof BG, Gillespie DL, Gloviczki ML, Lohr JM, McLafferty RB, Meissner MH, Murad MH, Padberg FT, Pappas PJ, Passman MA, Raffetto JD, Vasquez MA, Wakefield TW; Society for Vascular Surgery; American Venous Forum. The care of patients with varicose veins and associated chronic venous diseases: clinical practice guidelines of the Society for Vascular Surgery and the American Venous Forum. J Vasc Surg. 2011 May;53(5 Suppl):2S-48S. doi: 10.1016/j.jvs.2011.01.079. PMID 21536172
- [Background] Marsden G, Perry M, Kelley K, Davies AH; Guideline Development Group. Diagnosis and management of varicose veins in the legs: summary of NICE guidance. BMJ. 2013 Jul 24;347:f4279. doi: 10.1136/bmj.f4279. No abstract available. PMID 23884969
- [Background] Edwards AG, Baynham S, Lees T, Mitchell DC. Management of varicose veins: a survey of current practice by members of the Vascular Society of Great Britain and Ireland. Ann R Coll Surg Engl. 2009 Jan;91(1):77-80. doi: 10.1308/003588409X358953. Epub 2008 Nov 4. PMID 18990266
- [Background] Fonken LK, Weil ZM, Nelson RJ. Mice exposed to dim light at night exaggerate inflammatory responses to lipopolysaccharide. Brain Behav Immun. 2013 Nov;34:159-63. doi: 10.1016/j.bbi.2013.08.011. Epub 2013 Sep 6. PMID 24012645
- [Background] Elderman JH, Krasznai AG, Voogd AC, Hulsewe KW, Sikkink CJ. Role of compression stockings after endovenous laser therapy for primary varicosis. J Vasc Surg Venous Lymphat Disord. 2014 Jul;2(3):289-96. doi: 10.1016/j.jvsv.2014.01.003. Epub 2014 Feb 14. PMID 26993388
- [Background] Hamel-Desnos CM, Guias BJ, Desnos PR, Mesgard A. Foam sclerotherapy of the saphenous veins: randomised controlled trial with or without compression. Eur J Vasc Endovasc Surg. 2010 Apr;39(4):500-7. doi: 10.1016/j.ejvs.2009.11.027. Epub 2010 Jan 25. PMID 20097585
- [Background] Whiteley MS, Dos Santos SJ, Fernandez-Hart TJ, Lee CT, Li JM. Media Damage Following Detergent Sclerotherapy Appears to be Secondary to the Induction of Inflammation and Apoptosis: An Immunohistochemical Study Elucidating Previous Histological Observations. Eur J Vasc Endovasc Surg. 2016 Mar;51(3):421-8. doi: 10.1016/j.ejvs.2015.11.011. Epub 2016 Jan 17. PMID 26790396
- [Derived] Joyce DP, Walsh SR, Yap CJQ, Chong TT, Tang TY. Compression therapy following ClariVein(R) ablation therapy: a randomised controlled trial of COMpression Therapy Following MechanO-Chemical Ablation (COMMOCA). Trials. 2019 Dec 5;20(1):678. doi: 10.1186/s13063-019-3787-4. PMID 31806052